CLINICAL TRIAL: NCT00002440
Title: An Open-Label, Phase II Trial to Evaluate the Steady-State Pharmacokinetics, Safety, and Efficacy of 1592U89 in Combination With Selected HIV-1 Protease Inhibitors in Antiretroviral-Naive, HIV-1-Infected Patients.
Brief Title: A Study of 1592U89 in Combination With Protease Inhibitors in HIV-Infected Patients Who Have Never Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238J; CNAA2004
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-11

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Mutation; HIV-1 Reverse Transcriptase; HIV Protease; Reverse Transcriptase Inhibitors; Anti-HIV Agents; abacavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir; abacavir; amprenavir; Nelfinavir; Saquinavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir
Drug: Abacavir sulfate
Drug: Amprenavir
Drug: Nelfinavir mesylate
Drug: Saquinavir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give 1592U89 plus certain protease inhibitors (PIs) to HIV-infected patients who never have been treated with anti-HIV drugs. This study also examines how the body processes these drugs when they are given together.

DETAILED DESCRIPTION:
In this Phase II, open-label study patients (16 per treatment group) are randomized to receive 1592U89 in combination with one of five protease inhibitors: indinavir, saquinavir, ritonavir, nelfinavir, or 141W94 for up to 48 weeks.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Local treatment for Kaposi's sarcoma.
* GM-CSF, G-CSF or erythropoietin.

Patients must have:

* HIV-1 infection documented by a licensed HIV-1 antibody ELISA and confirmed by Western blot detection of HIV-1 antibody or a positive HIV-1 blood culture.
* CD4+ cell count >= 100 cells/mm3 within 14 days of study drug administration.
* HIV-1 RNA >= 5,000 copies/ml within 14 days of study drug administration.
* No active or ongoing AIDS-defining opportunistic infection or disease.
* Signed, informed consent from parent or legal guardian for patients less than 18 years of age.

Prior Medication:

Allowed:

Local treatment for Kaposi's sarcoma.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malabsorption syndrome, or other gastrointestinal dysfunction, that might interfere with drug absorption or render the patient unable to take oral medication.
* Life-threatening infection or other serious medical condition that may compromise a patient's safety.

Concurrent Medication:

Excluded:

* Other investigational agents. NOTE:
* Those available through Treatment IND or expanded access programs are evaluated individually.
* Chemotherapeutic agents for the initial 24 weeks of study (except local treatment for Kaposi's sarcoma).
* Agents with documented anti-HIV activity in vitro.
* Foscarnet.
* Immunomodulating agents such as systemic corticosteroids, interleukins, thalidomide, anti-cytokine agents or interferons.
* Antioxidants.

Concurrent Treatment:

Excluded:

Radiation therapy within the first 24 weeks of study.

Patients with the following prior conditions are excluded:

* History of clinically relevant pancreatitis or hepatitis within the last 6 months.
* Participation in an investigational HIV-1 vaccine trial.

Prior Medication:

Excluded:

* Antiretroviral therapy, including reverse transcriptase inhibitor and protease inhibitor therapy.
* Cytotoxic chemotherapeutic agents within 30 days of study drug administration.
* HIV-1 vaccine dose within the 3 months prior to study drug administration.
* Immunomodulating agents, such as systemic corticosteroids, interleukins or interferons within 30 days of study drug administration.

Prior Treatment:

Excluded:

Radiation therapy within 30 days of study drug administration. Alcohol or illicit drug use that may interfere with patient compliance.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - UCSD Treatment Ctr, San Diego, California
  - Yale U / New Haven Med Ctr / AIDS Clinical Trials Unit, New Haven, Connecticut
  - Kansas City AIDS Research Consortium, Kansas City, Missouri
  - NYU Med Ctr / Dept of Medicine / AIDS Clinical Trial, New York, New York
  - Carolinas Med Ctr, Charlotte, North Carolina
  - Case Western Reserve Univ / AIDS Clinical Trials Unit, Cleveland, Ohio
  - Univ of Pittsburgh Med Ctr, Pittsburgh, Pennsylvania
  - Vanderbilt Univ Med Ctr, Nashville, Tennessee